CLINICAL TRIAL: NCT00666198
Title: Special Investigation For Long-term Use Of Revatio (Regulatory Post Marketing Commitment Plan)
Brief Title: Special Investigation For Long-Term Use Of Sildenafil (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481263
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SILDENAFIL: Patients taking SILDENAFIL.
  Interventions: Drug: SILDENAFIL

INTERVENTIONS:
Drug: SILDENAFIL — Revatio® Tablets 20 mg Dosage, Frequency: According to Japanese LPD, "For oral use, the adult dose is 20 mg three times a day".
  Duration: According to the protocol of A1481263, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 3 years after the first administration.

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first SILDENAFIL(Revatio) should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered SILDENAFIL(Revatio) in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered SILDENAFIL(Revatio).

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A1481263 prescribes the SILDENAFIL(Revatio).
Sampling Method: Probability Sample
Enrollment: 3337 (Actual)
Dates: Start 2008-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481263&StudyName=Special%20Investigation%20For%20Long-Term%20Use%20Of%20Sildenafil%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Revatio (Sildenafil Citrate): Participants who received Revaio (Sildenafil citrate) as indicated in the approved local product document were observed for a period of 3 years. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Revatio (Sildenafil Citrate)
Started | 3337
Completed | 3304
Not Completed | 33
Not completed — Protocol Violation | 10
Not completed — No Visit After First Day of Treatment | 13
Not completed — Safety Not Assessable | 6
Not completed — No Drug Administration | 4

BASELINE CHARACTERISTICS:
Population: A total of 3304 participants received sildenafil citrate at least once in this study. Of the 3304 participants, 33 participants were excluded from the baseline analysis due to following reasons: protocol violation, no visit after first day of treatment, safety not assessable and no drug administration.
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Age, Customized [Number; unit: Participants]
  ˂65 years | 2406
  ≥65 years | 898
Age, Customized [Number; unit: Participants]
  ˂15 years | 1050
  ≥15 years | 2254
Sex/Gender, Customized [Number; unit: Participants]
  Female | 2057
  Male | 1247
Disease Type [Number; unit: Participants] — Categorization of PAH in the study. * indicates "Associated Pulmonary Arterial Hypertension (APAH)". ** refers to "Pulmonary Veno Occlusive Disease/Pulmonary Capillary Hemangiomatosis".
  Participants
    Idiopathic/Familial PAH (IPAH/FPAH) | 745
    Collagen Vascular Disease* | 666
    Congenital Systemic to Pulmonary Shunts* | 985
    PVOD/PCH** | 44
    Persistent PH of the Newborn (PPHN) | 59
    Other PAH (Portal Hypertention/HIV Infection etc.) | 139
    Other Than PAH | 665
    Unknown | 1
WHO Functional Classification of PAH [Number; unit: Participants] — This system grades PAH severity according to the functional status of the patient. The grades range from Functional Class (FC) I, where the patient's disease does not affect their day-to-day activities, to FC IV, where patients are severely functionally impaired, even at rest. This functional classification system links symptoms with activity limitations, and allows clinicians to quickly predict disease progression and prognosis, as well as the need for specific treatment regimens, irrespective of the underlying etiology of PAH.
  Participants
    Class I | 344
    Class II | 1012
    Class III | 1279
    Class IV | 545
    Not Classified | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to sildenafil citrate was assessed by the physician/investigator.
Time Frame: 3 years
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received sildenafil citrate at least once.
Measure: Number; unit: Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Participants
  Treatment-Related Adverse Event | 448
  Treatment-Related Serious Adverse Event | 101

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to sildenafil citrate was assessed by the physician/investigator.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Participants | 196

3. Primary Outcome: Number of Paritcipants With Treatment-Related Adverse Events by Age
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. Relatedness to sildenafil citrate was assessed by the physician/investigator. Participants with treatment related adverse events were counted by age to assess whether it was risk factor for the treatment related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Paritcipants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Paritcipants
  ˂15 years (n=1050) | 57
  ≥15 years (n=2254) | 391

4. Primary Outcome: Number of Paritcipants With Treatment-Related Adverse Events by Gender
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. Relatedness to sildenafil citrate was assessed by the physician/investigator. Participants with treatment related adverse events were counted by gender to assess whether it was risk factor for the treatment related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Paritcipants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Paritcipants
  Female (n=2057) | 323
  Male (n=1247) | 125

5. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Disease Type
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. Relatedness to sildenafil citrate was assessed by the physician/investigator. Participants with treatment related adverse events were counted by disease type to assess whether it was risk factor for the treatment related adverse events.
  * indicates "Associated Pulmonary Arterial Hypertension (APAH)". ** refers to "Pulmonary Veno Occlusive Disease/Pulmonary Capillary Hemangiomatosis".
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Participants
  Idiopathic/Familial PAH(IPAH/FPAH) (n=745) | 116
  Collagen Vascular Disease* (n=666) | 136
  Congenital Systemic to Pulmonary Shunts* (n=985) | 66
  PVOD/PCH** (n=44) | 4
  Persistent PH of the Newborn (PPHN) (n=59) | 3
  Other PAH (n=139) | 25
  Other Than PAH (n=665) | 98
  Unkown (n=1) | 0

6. Primary Outcome: Number of Participants With Treatmnt-Related Adverse Events by WHO Functional Classification of Severity
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sildenafil citrate in a participant who received sildenafil citrate. Relatedness to sildenafil citrate was assessed by the physician/investigator. Participants with treatment related adverse events were counted by severity (WHO functional classification for PAH range;This system grades PAH severity according to the functional status of the patient. The grades range from Functional Class (FC) I, where the patient's disease does not affect their day-to-day activities, to FC IV, where patients are severely functionally impaired, even at rest. This functional classification system links symptoms with activity limitations, and allows clinicians to quickly predict disease progression and prognosis, as well as the need for specific treatment regimens, irrespective of the underlying etiology of PAH) to assess whether it was risk factor for the treatment related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3304
Participants
  Class I (n=344) | 34
  Class II (n=1012) | 127
  Class III (n=1279) | 204
  Class IV (n=545) | 63
  Not Classified (n=124) | 20

7. Primary Outcome: Clinical Efficacy Rate by Age
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of sildenafil citrate was assessed as "effective," "ineffective" or "unassessable" by the physician/investigator. Overall effectiveness of sildenafil citrate was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as echocardiogram. Participants achieved clinical effectiveness by age were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 3 years
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician/investigator based upon change in clinical symptoms and laboratory findings) at least once. Participants with observed effectiveness data were included in table.
Measure: Number; unit: Percentage of Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3301
Percentage of Participants
  ˂15 years (n=1049) | 72.0
  ≥15 years (n=2252) | 62.0

8. Primary Outcome: Clinical Efficacy Rate by Gender
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of sildenafil citrate was assessed as "effective," "ineffective" or "unassessable" by the physician/investigator. Overall effectiveness of sildenafil citrate was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as echocardiogram. Participants achieved clinical effectiveness by gender were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 3 years
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3301
Percentage of Participants
  Female (n=2054) | 65.9
  Male (n=1247) | 64.0

9. Primary Outcome: Clinical Efficacy Rate by Disease Type
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of sildenafil citrate was assessed as "effective," "ineffective" or "unassessable" by the physician/investigator. Overall effectiveness of sildenafil citrate was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as echocardiogram. Participants achieved clinical effectiveness by disease type were counted to assess whether it contributes to the clinical effectiveness.
  * indicates "Associated Pulmonary Arterial Hypertension (APAH)". ** refers to "Pulmonary Veno Occlusive Disease/Pulmonary Capillary Hemangiomatosis".
Time Frame: 3 years
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3301
Percentage of Participants
  Idiopathic/Familial PAH(IPAH/FPAH) (n=743) | 67.6
  Collagen Vascular Disease* (n=666) | 61.6
  Congenital Systemic to Pulmonary Shunts* (n=984) | 72.9
  PVOD/PCH** (n=44) | 40.9
  Persistent PH of the Newborn (PPHN) (n=59) | 55.9
  Other PAH (n=139) | 67.6
  Other Than PAH (n=665) | 56.5
  Unknown (n=1) | 100.0

10. Primary Outcome: Clinical Efficacy Rate by WHO Functional Classificaton of Severity
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of sildenafil citrate was assessed as "effective," "ineffective" or "unassessable" by the physician/investigator. Overall effectiveness of sildenafil citrate was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as echocardiogram. Participants achieved clinical effectiveness by severity (WHO functional classification of PAH;The grades range from Functional Class (FC) I, where the patient's disease does not affect their day-to-day activities, to FC IV, where patients are severely functionally impaired, even at rest. This functional classification system links) were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 3 years
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Revatio (Sildenafil Citrate)
Number analyzed (Participants) | 3301
Percentage of Participants
  Class I (n=344) | 76.2
  Class II (n=1010) | 70.5
  Class III (n=1279) | 64.2
  Class IV (n=544) | 52.4
  Not Classified (n=124) | 57.3

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Revatio (Sildenafil Citrate)
Serious Adverse Events (participants affected / at risk) | 982/3304
Other Adverse Events (participants affected / at risk) | 509/3304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revatio (Sildenafil Citrate) (N=3304)
Appendicitis (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Campylobacter gastroenteritis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 19
Bronchiolitis (Infections and infestations) | 1
Brain abscess (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 4
Disseminated tuberculosis (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis adenovirus (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 2
Hepatitis A (Infections and infestations) | 1
Infection (Infections and infestations) | 6
Influenza (Infections and infestations) | 7
Laryngitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Meningitis (Infections and infestations) | 4
Meningitis aseptic (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Oesophageal candidiasis (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 86
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 2
Pneumonia staphylococcal (Infections and infestations) | 2
Pseudomembranous colitis (Infections and infestations) | 2
Pulmonary mycosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 3
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 20
Septic embolus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Infusion site infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 3
Catheter site infection (Infections and infestations) | 6
Phlebitis infective (Infections and infestations) | 1
Wound abscess (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Klebsiella bacteraemia (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 10
Serratia infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Puncture site infection (Infections and infestations) | 3
Device related infection (Infections and infestations) | 26
Device related sepsis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3
Candida infection (Infections and infestations) | 1
Varicella zoster pneumonia (Infections and infestations) | 1
Cholangitis infective (Infections and infestations) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to gallbladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
POEMS syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Abnormal clotting factor (Blood and lymphatic system disorders) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 19
Anaemia neonatal (Blood and lymphatic system disorders) | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 10
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 3
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Thrombocytosis (Blood and lymphatic system disorders) | 1
Allergic granulomatous angiitis (Immune system disorders) | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 2
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Aggression (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 2
Self injurious behaviour (Psychiatric disorders) | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Altered state of consciousness (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 8
Cerebral infarction (Nervous system disorders) | 9
Clonic convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 2
Febrile convulsion (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 5
Intracranial pressure increased (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 3
Neuropsychiatric lupus (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Seizure anoxic (Nervous system disorders) | 1
Spastic paralysis (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Visual impairment (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 8
Atrial flutter (Cardiac disorders) | 5
Atrial tachycardia (Cardiac disorders) | 4
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 2
Bradyarrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 14
Cardiac failure (Cardiac disorders) | 156
Cardiac failure acute (Cardiac disorders) | 8
Cardiac failure chronic (Cardiac disorders) | 16
Cardiac failure congestive (Cardiac disorders) | 18
Cardiac tamponade (Cardiac disorders) | 1
Cardiac valve disease (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 12
Cardiovascular insufficiency (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 6
Left ventricular dysfunction (Cardiac disorders) | 1
Low cardiac output syndrome (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 5
Pericardial effusion (Cardiac disorders) | 2
Pericarditis constrictive (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 44
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 3
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 4
Tricuspid valve incompetence (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 2
Ventricular fibrillation (Cardiac disorders) | 5
Ventricular tachycardia (Cardiac disorders) | 6
Arteriovenous fistula (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 13
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 10
Kawasaki's disease (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Shock (Vascular disorders) | 8
Shock haemorrhagic (Vascular disorders) | 2
Vena cava thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diffuse panbronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 67
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 17
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 17
Pulmonary haemosiderosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 112
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary vein occlusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 46
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 6
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 3
Faeces discoloured (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7
Gastrointestinal hypomotility (Gastrointestinal disorders) | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 5
Ileus paralytic (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophageal fistula (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Portal venous gas (Gastrointestinal disorders) | 1
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 5
Rectal polyp (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Biliary cirrhosis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 7
Hepatic congestion (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 9
Hepatic function abnormal (Hepatobiliary disorders) | 25
Hepatitis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 4
Portal hypertension (Hepatobiliary disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subepidermal (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 12
Acute prerenal failure (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 4
Diabetic nephropathy (Renal and urinary disorders) | 1
Prerenal failure (Renal and urinary disorders) | 3
Renal disorder (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 15
Renal impairment (Renal and urinary disorders) | 8
Scleroderma renal crisis (Renal and urinary disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 2
Atrial septal defect (Congenital, familial and genetic disorders) | 2
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 1
Congenital mitral valve stenosis (Congenital, familial and genetic disorders) | 1
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Interruption of aortic arch (Congenital, familial and genetic disorders) | 1
Mitochondrial myopathy (Congenital, familial and genetic disorders) | 1
Persistent foetal circulation (Congenital, familial and genetic disorders) | 4
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 2
Pulmonary artery atresia (Congenital, familial and genetic disorders) | 2
Pulmonary hypoplasia (Congenital, familial and genetic disorders) | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1
Catheter site erythema (General disorders) | 1
Catheter site induration (General disorders) | 1
Catheter site swelling (General disorders) | 1
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 3
Death (General disorders) | 24
Device breakage (General disorders) | 2
Device connection issue (General disorders) | 1
Device damage (General disorders) | 3
Device pacing issue (General disorders) | 1
Disease progression (General disorders) | 13
Food interaction (General disorders) | 1
General physical health deterioration (General disorders) | 1
Generalised oedema (General disorders) | 3
Inflammation (General disorders) | 1
Malaise (General disorders) | 2
Multi-organ failure (General disorders) | 17
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 7
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 4
Sudden infant death syndrome (General disorders) | 1
Thirst (General disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood glucose abnormal (Investigations) | 1
Blood pressure decreased (Investigations) | 9
Blood pressure increased (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 7
Carbon dioxide increased (Investigations) | 1
Cardiac output decreased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 1
Computerised tomogram thorax abnormal (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
International normalised ratio increased (Investigations) | 3
Liver function test abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 12
Pulmonary arterial pressure increased (Investigations) | 2
Serum ferritin increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight increased (Investigations) | 1
Arterial injury (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Stab wound (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 7
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Catheter removal (Surgical and medical procedures) | 1
Lung transplant (Surgical and medical procedures) | 1
Skin operation (Surgical and medical procedures) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Revatio (Sildenafil Citrate) (N=3304)
Bronchitis (Infections and infestations) | 82
Anaemia (Blood and lymphatic system disorders) | 74
Headache (Nervous system disorders) | 136
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 71
Diarrhoea (Gastrointestinal disorders) | 79
Hepatic function abnormal (Hepatobiliary disorders) | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.